CLINICAL TRIAL: NCT01478451
Title: Danish: Integreret Motion på Arbejdspladsen (IRMA) English: Implementation of Exercise at the Workplace
Brief Title: Acute Effect of Massage and Exercise on Muscle Tenderness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Responsible Party: Principal Investigator, Lars L. Andersen, Principal Investigator, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IRMA02
Record Dates: First submitted 2011-10-28; First posted 2011-11-23 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Musculoskeletal Disorders
Keywords: DOMS
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Exercise; Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Massage (Experimental): massage will be provided for 10 minutes at the left or right trapezius (randomized)
  Interventions: Other: Massage
- Exercise (Experimental): exercise (shoulder shrugs with elastic resistance) will be performed for 10 minutes at the left or right trapezius (randomized)
  Interventions: Behavioral: Exercise
- Control (No Intervention): control shoulder (randomized)

INTERVENTIONS:
Behavioral: Exercise — Exercise will be performed for 10 minutes at the left or right trapezius (randomized)
  Arms: Exercise
Other: Massage — massage will be provided for 10 minutes at the left or right trapezius (randomized)
  Arms: Massage

SUMMARY:
Many people experience pain, tenderness and soreness of joint and muscles, both in sport and working life. Pain killers can provide acute relief of pain, but may not be a feasible solution for all people. Here the investigators examine the acute effect of massage and exercise on induced muscle tenderness (delayed onset muscular soreness).

ELIGIBILITY:
Inclusion Criteria:

* working age adults

Exclusion Criteria:

* blood pressure above 160/100
* disease of the cervical spine

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Perceived tenderness of the trapezius muscle on a numerical rating scale of 0-10 | change from before to after the acute intervention (average of 0, 10, 20 and 60 min after the intervention)
  Perceived tenderness where 0 is no tenderness and 10 is worst imaginable tenderness
Pressure pain threshold of the trapezius muscle | change from before to after the acute intervention (average of 0, 10, 20 and 60 min after the intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Lars L Andersen, PhD, Principal Investigator — Senior Researcher
Locations (1):
- National Research Centre for the Working Environment, Copenhagen, Denmark

REFERENCES:
- [Derived] Andersen LL, Jay K, Andersen CH, Jakobsen MD, Sundstrup E, Topp R, Behm DG. Acute effects of massage or active exercise in relieving muscle soreness: randomized controlled trial. J Strength Cond Res. 2013 Dec;27(12):3352-9. doi: 10.1519/JSC.0b013e3182908610. PMID 23524365
- See also: Related Info — http://arbejdsmiljoforskning.dk